CLINICAL TRIAL: NCT01403935
Title: Sepsis Institutional Registry in Hospital Italiano de Buenos Aires
Acronym: SIR
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1172
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Death; Severe Sepsis
MeSH Terms: conditions — Death; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create an institutional registry of sepsis through a prospective survey based on epidemiological data, risk factors, diagnosis, prognosis, treatment, monitoring and survival.

DETAILED DESCRIPTION:
The main goal is to describe the occurrence of sepsis and the characteristics of clinical presentation, evolution and predisposing factors within the population of the Hospital Italiano de Buenos Aires.

ELIGIBILITY:
Inclusion Criteria:

1. Over 17 years
2. Two or more sirs criteria
3. Active infection

Exclusion Criteria:

1. Refusal to register or to the informed consent process
2. Ambulatory patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 7472 (Actual)
Dates: Start 2007-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
clinical features, mortality | Clinical characteristics are evaluated during the acute event and in-hospital mortality and annual monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Gascon 450, Buenos Aires, Argentina